CLINICAL TRIAL: NCT02594137
Title: A Randomized Controlled Study Comparing 2 Surgical Techniques for Decompressive Craniectomy: With Watertight Duraplasty Versus Without Watertight Duraplasty.
Brief Title: A Comparison Between Two Techniques for Performing Decompressive Craniectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital of the Restoration, Recife (Other)
Responsible Party: Principal Investigator, Eduardo Vieira de Carvalho Junior, Professor in Residence of Neurological Surgery, Hospital of the Restoration, Recife
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0115.0.102.000-11
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Brain Edema; Craniocerebral Trauma; Infarction, Middle Cerebral Artery
Keywords: Decompressive craniectomy; Brain Edema
MeSH Terms: conditions — Brain Edema; Craniocerebral Trauma; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Watertight Duraplasty (Experimental): After standard craniectomy (12x15cm) and dural opening, the "intervention", which is to not perform watertight duraplasty is carried out. The exposed brain parenchyma is covered with Surgicel. Usual closure is then performed.
  Interventions: Procedure: Without watertight duraplasty
- With Watertight Duraplasty (No Intervention): After standard craniectomy (12x15cm) and dural opening, watertight duraplasty with pericranium or an artificial graft is performed. Usual closure is then performed. This kind of duraplasty is performed by most neurosurgeons and this group will be used as a control.

INTERVENTIONS:
Procedure: Without watertight duraplasty — After standard craniectomy and dural opening, provided there is no brain contusions or hematomas requiring surgical evacuation, no watertight duraplasty is performed. The dura is left opened and the brain parenchyma is covered with Surgicel. Usual closure is then performed.
  Arms: Without Watertight Duraplasty

SUMMARY:
The purpose of this study is to compare two surgical techniques for a neurosurgical procedure used to treat cerebral edema (decompressive craniectomy): with watertight duraplasty vs. without watertight duraplasty (rapid closure decompressive craniectomy).

DETAILED DESCRIPTION:
After clinical indication for unilateral decompressive craniectomy (DC), patients were randomized by numbered envelopes into 2 groups: with watertight duraplasty (control group) vs. without watertight duraplasty / rapid closure DC (test group). In all cases, a large trauma flap (i.e. large reverse question mark starting from the tragus and extending to the midline) was performed. Skin, galea and muscle layers were elevated according to surgeon preference. Thus a wide (at least 12x15cm) craniotomy was performed and the temporal bone was removed until flush with the middle fossa floor. After dural opening, watertight duraplasty with pericranium or an artificial graft (at surgeon's discretion) was performed in the control group, while no watertight duraplasty was performed in the test group, and exposed brain parenchyma was covered with Surgicel®. Usual closure was then performed. Patients were then monitored daily by evaluators blinded to the randomization (control or test group) from the date of surgery until hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Neurotrauma Service of the Hospital of Restoration from January 2012 to December 2013, age range 18 to 60 years old and with clinical indication for decompressive craniectomy.

Exclusion Criteria:

* Indication for bifrontal decompressive craniectomy.
* Indication for Posterior Fossa decompressive craniectomy
* Patients with intra-axial contusions or hematomas requiring surgical evacuation in which case injury to the arachnoid could lead to an increased risk of cerebrospinal fluid leak

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Surgical Complications | From surgical procedure until hospital discharge or death (maximum of 90 days)
  Cerebrospinal Fluid Leaks, Wound Infection, Brain Abscess, Subgaleal Fluid Collections)

SECONDARY OUTCOMES:
Clinical Outcome (Analyzed by the Glasgow Outcome Scale) | From surgical procedure until hospital discharge or death (maximum of 90 days)
Hospital Costs | From surgical procedure until hospital discharge or death (maximum of 90 days)
Surgical Time | From skin incision until closure is completed (maximum of 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo V Carvalho Junior, MD, Principal Investigator — Hospital of the Restoration

REFERENCES:
- [Background] Guresir E, Vatter H, Schuss P, Oszvald A, Raabe A, Seifert V, Beck J. Rapid closure technique in decompressive craniectomy. J Neurosurg. 2011 Apr;114(4):954-60. doi: 10.3171/2009.12.JNS091065. Epub 2010 Jan 29. PMID 20113157
- [Background] Barth M, Tuettenberg J, Thome C, Weiss C, Vajkoczy P, Schmiedek P. Watertight dural closure: is it necessary? A prospective randomized trial in patients with supratentorial craniotomies. Neurosurgery. 2008 Oct;63(4 Suppl 2):352-8; discussion 358. doi: 10.1227/01.NEU.0000310696.52302.99. PMID 18981842
- [Background] Sade B, Oya S, Lee JH. Non-watertight dural reconstruction in meningioma surgery: results in 439 consecutive patients and a review of the literature. Clinical article. J Neurosurg. 2011 Mar;114(3):714-8. doi: 10.3171/2010.7.JNS10460. Epub 2010 Aug 13. PMID 20707618
- [Background] Ragel BT, Klimo P Jr, Martin JE, Teff RJ, Bakken HE, Armonda RA. Wartime decompressive craniectomy: technique and lessons learned. Neurosurg Focus. 2010 May;28(5):E2. doi: 10.3171/2010.3.FOCUS1028. PMID 20568936
- [Background] Kolias AG, Kirkpatrick PJ, Hutchinson PJ. Decompressive craniectomy: past, present and future. Nat Rev Neurol. 2013 Jul;9(7):405-15. doi: 10.1038/nrneurol.2013.106. Epub 2013 Jun 11. PMID 23752906
- [Derived] Vieira E, Guimaraes TC, Faquini IV, Silva JL, Saboia T, Andrade RVCL, Gemir TL, Neri VC, Almeida NS, Azevedo-Filho HRC. Randomized controlled study comparing 2 surgical techniques for decompressive craniectomy: with watertight duraplasty and without watertight duraplasty. J Neurosurg. 2018 Oct;129(4):1017-1023. doi: 10.3171/2017.4.JNS152954. Epub 2017 Nov 17. PMID 29148904